CLINICAL TRIAL: NCT04741230
Title: Prospective, Investigator Initiated Feasibility Study to Evaluate the Safety, and Indicative Effectiveness of Gebauer™ Lenticules in Patients Suffering From Severe Keratoconus or Post LASIK Ectasia
Brief Title: Investigator Initiated, Prospective Study of Xenia Corneal Lenticule
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Collaborators: Gebauer Company (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019OPH108
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Keratoconus; Post-Laser Retinal Condition
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gebauer Lenticule (Experimental): Gebauer Lenticule implant device
  Interventions: Device: Gebauer Lenticule

INTERVENTIONS:
Device: Gebauer Lenticule — The Gebauer™ Lenticule corneal implant device is a custom-made device intended for patients suffering from keratoconus or post-LASIK ectasia. The device is expected to reinforce and stabilize the patient's cornea, so that a more consistent refraction is induced and a penetrating human cornea donor transplantation may be avoided or postponed.

SUMMARY:
Cornea ectatic conditions such as keratoconus and post-LASIK (Laser In situ Keratomileusis) ectasia are disorders of the eye that are notorious for its uncontrolled progression over time, leading to loss of vision. There are valuable treatment options for controlling disease progression in mild to moderate stages of such disease. However in advanced cases and / or when contact lenses cannot be worn, surgery remains the only treatment option to rehabilitate vision. Most treatment options are highly invasive and represent significant risks. This study evaluates a novel corneal implant, Gebauer™ Lenticule to treat severe keratoconus or post-LASIK ectasia. This implant is derived from porcine collagen and intended for intra-stromal insertion. The Gebauer™ Lenticule is expected to improve the stability of the cornea while not impairing the vision. The procedure is an additive procedure after other treatment options have been exhausted. The procedure is reversible with removal of the implant (in the unexpected case of an adverse reaction), and vision may be restored to baseline.

The purpose of this study is to evaluate how well the implant is tolerated, it's safety profile, and how effective this new treatment option is in the treatment of keratoconus or post-LASIK ectasia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe keratoconus in patients who would prefer to avoid corneal transplant surgery / penetrating keratoplasty OR
* Diagnosis of severe post-LASIK Ectasia in patients who would prefer to avoid corneal transplant surgery / penetrating keratoplasty
* In terms of general health, patients must be free of diagnosed terminal illnesses (life expectancy of greater than or equal to 2 years).
* Patients must be aged 18 years or over and less than 80 years old
* Patients' contact lenses must have been removed at least one-week prior to surgery for soft lenses and two weeks prior to surgery for hard lenses
* Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed
* Patient must be able and willing to complete all study visits and comply with the study-specific requirements

Exclusion Criteria:

* History or presence of any ocular pathologies that may interfere with the planned surgical treatment, including corneal epithelial problems
* Previous corneal transplantation or corneal implant in the designated eye
* Cataract with anticipated surgical intervention (IOL implantation) within 2 years
* Active inflammation and/or infection of the eye or the eye lid
* Patients with Intra Ocular Pressure (IOP) <10 mmHg or >21 mmHg
* Professionally diagnosed and currently treated autoimmune diseases
* Current strong symptoms of any allergy
* History of major organ transplantation and/or current continuing immunosuppressive treatment
* History of blood transfusion within the last 12 months
* Subject who is currently participating or has participated in another investigational clinical study within the past 60 days Pregnancy and lactation

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Immunological rejection by ophthalmic examination of Intraocular pressure, Best corrected visual acuity, Corneal and Lenticule transparency, Inflammation | 6 months
  Signs of immunological rejection during the post implantation observation period
Treatment-related adverse events. | 6 months
  The frequency and severity of all treatment-related adverse events, during implantation of the Gebauer™ Lenticule and throughout the post implantation observation period.
Changes in corneal topography (central K-reading results) | 6 months
  Changes in corneal topography (central K-reading results): at baseline vs. post implantation observation period
Central corneal thickness | 6 months
  Changes in central corneal thickness at baseline vs. post implantation corneal thickness (cornea plus lenticule)

CONTACTS AND LOCATIONS:
Overall Officials: B Ilango, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands, United Kingdom